CLINICAL TRIAL: NCT00062998
Title: Free-Living Physical Activity and Energy Expenditure
Status: Completed | Type: Observational
Sponsor: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Other Study IDs: R03 (DK62152) (completed 2006); R03DK062152 (NIH)
Record Dates: First submitted 2003-06-18; First posted 2003-06-19 (Estimated); Last update posted 2010-03-18 (Estimated); Status verified 2010-03

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Time Perspective: Prospective

SUMMARY:
We have recently validated a new device for measurement of physical activity and found it to detect type, duration and intensity of many types of physical activity at better than 98% accuracy. After further validating this device to determine if it can also accurately assess energy expenditure, we will use it to collect cross-sectional data on free-living physical activity and energy expenditure in adolescent girls.

ELIGIBILITY:
Study3: healthy lean and obese adults, at least 18 years of age.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 15

CONTACTS AND LOCATIONS:
Locations (1):
- St. Luke's-Roosevelt Hospital Center, New York, New York, United States